CLINICAL TRIAL: NCT06831201
Title: Effect of Different Proprioceptive Neuromuscular Facilitation Techniques Versus Flow Trigger Sensitivity on Weaning Off Mechanical Ventilation
Acronym: PNF techniques
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, yasmin sabry abdelnabi hassan, sponsor-investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FPTBSUREC/0103/241124
Record Dates: First submitted 2025-01-27; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Failure
Keywords: Mechanical ventilation; Flow triggering senstivity; Different proprioceptive techniques
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Trigger sensitivity training (Experimental): *Training will be based on decreasing the trigger sensitivity gradually in order to increase muscle endurance.
  Interventions: Device: Flow trigger sensitivity group
- Active proprioceptive facilitation technique (active PNF technique) (Active Comparator): PNF techniques included one session of physiotherapy including four 90-second manual stimulations each (upper ribs, lower ribs, sternum, and diaphragm). First, patients in this group will be treated with the rhythmic initiation technique (RIT) derived from the PNF concept. This technique facilitates the correct movement pattern, improves coordination and movement awareness of the chest wall.
  Second, patients in this group will be treated with the initial stretch technique (IST), a technique also originating from the PNF concept (named also as: repeated stretch from beginning of range or repeated initial stretch).This technique facilitates the initiation of inhalation.
  Interventions: Procedure: Active proprioceptive facilitation technique ( active PNF) technique
- Passive proprioceptive facilitation technique ( passive PNF technique ) (Active Comparator): Passive PNF methods are those involving the application of external proprioceptive and tactile stimuli producing reactions to reflex respiratory movement that appear to change breathing frequency and depth by this mechanism control and coordination movements of thoracic cage were facilitated and there is improvement in chest expansion and compliance. those methods include Perioral Pressure, Expanded epigastric movement ,Intercostal Stretch, Thoracic Vertebral Pressure, Co-contraction of the Abdomen ,Moderate Manual Pressure, Anterior Stretch-Lifting of the Posterior Basal Area (Basal Lift).
  Interventions: Procedure: Passive proprioceptive facilitation technique ( passive PNF) technique

INTERVENTIONS:
Device: Flow trigger sensitivity group — 1. Pressure support ventilation will be titrated at a level sufficient to achieve a respiratory rate of 20-30 breath/min and tidal volume 4-6 ml/kg. Pressure support will be reduced by 2 cm H2O every hour to reach pressure support 8 cm H2O. Two exercise sessions will be performed, at 9 AM and 5 PM. Training will be based on decreasing the trigger sensitivity gradually in order to increase muscle endurance. The trigger sensitivity will be adjusted to 20% of the first recorded MIP at the start of training (In the first session), inspiratory muscle training (IMT) will be limited to 5 min; afterwards the duration will be increased by 5 min at every session until it reach 30 min. If a patient tolerates 30 min of IMT, The next session will be performed with increasing trigger sensitivity by 10% of the initial MIP. Patients who could not tolerate IMT with 20% of MIP for 5 min were trained with 10% of MIP. Training consists of 5 to 6 sets of repetitions through the trainer.
  Arms: Trigger sensitivity training
Procedure: Active proprioceptive facilitation technique ( active PNF) technique — 1. patients in this group treated with the rhythmic initiation technique derived from the PNF concept. The RIT will be applied in four manual positions of the therapist's hands: The upper and lower chest wall, the sternum and below the rib cage, so that the patient can learn the correct breathing pattern. Verbal commands will be also used by the PT to reinforce the manual stimulation with each pattern/exercise being performed 10 times.
  2. patients treated with the initial stretch technique ,This technique facilitates the initiation of inhalation. The IST was applied to help the patient to initiate the inhalation phase, increase the force developed by the inspiratory muscle, and to enhance the active range of motion of the chest wall and the diaphragm. At the final stage of exhalation, when inspiratory muscles will be elongated optimally, the stretch reflex will be initiated by applying a quick tap to elicit a strong and active inspiratory muscle contraction
  Arms: Active proprioceptive facilitation technique (active PNF technique)
Procedure: Passive proprioceptive facilitation technique ( passive PNF) technique — Perioral pressure is provided by applying pressure with the therapist's finger on the top lip between the nose and lip. The pressure is maintained for the length of time that the therapist wishes the patient to breathe in the activated pattern.
  Intercostal stretch is provided by applying pressure to the upper border of a rib in order to stretch the intercostal muscle in a downward(not inward) direction. The stretch position is then maintained while the patient continues to breathe in his/her usual manner.
  vertebral pressure high - manual pressure applied to thoracic vertebrae in the region T2 - T5.
  vertebral pressure low - manual pressure applied to thoracic vertebrae in the region T9 - T10.
  Co-contraction of the Abdomen Provided by the therapist by pressing adequate pressure on the lower ribs and pelvis on the same side, so that pressure is applied at right angles to the patient.
  Moderate Manual Pressure of the open hand(s) is maintained over the area in which expansion is desired
  Arms: Passive proprioceptive facilitation technique ( passive PNF technique )

SUMMARY:
Weaning is a critical stage in respiratory care, requiring strategies to optimize breathing muscle function and reduce patient dependence on ventilatory support.

PNF Techniques: These techniques are traditionally used to improve muscle strength and coordination. When applied to respiratory therapy, PNF can enhance diaphragmatic strength, improve chest wall mobility, and promote effective breathing patterns, potentially accelerating the weaning process.

Flow Trigger Sensitivity: This approach focuses on fine-tuning ventilator settings to ensure minimal patient effort in initiating breaths. By improving patient-ventilator synchronization, it reduces respiratory muscle fatigue and supports efficient weaning.

The study likely compares the two approaches in terms of weaning success rates, duration, and respiratory muscle performance. It may conclude that combining PNF techniques with optimized ventilator settings can improve weaning outcomes by enhancing respiratory muscle functionality and reducing mechanical ventilation dependency.

DETAILED DESCRIPTION:
PURPOSE The main aim of this study is to compare the effect of Different proprioceptive neuromuscular facilitation techniques versus Flow Trigger Sensitivity On Weaning Off Mechanical Ventilation BACKGROUND Respiratory failure occurs when the respiratory system fails adequately to oxygenate or eliminate carbon dioxide from the blood. Under such circumstances, mechanical ventilation is used to meet these demands artificially. When the precipitating cause of respiratory failure is corrected, most patients can easily resume spontaneous breathing and do not require any elaborate "weaning" techniques. In a few cases, however, especially when the precipitating cause cannot be completely corrected or when the complications of mechanical ventilation have aggravated respiratory failure, the patient cannot readily resume the work of breathing. In such cases, gradual weaning can usually allow mechanical ventilation to be discontinued safely and without excessive discomfort. Sometimes, unfortunately, the response to gradual weaning is poor; these patients continue to present a challenge to pulmonary and critical care physicians .

Mechanical ventilation (MV) supports breathing in critically ill patients in the setting of intensive care unit (ICU). Although indispensable, MV has been implicated in the dysfunction of the diaphragm and respiratory muscle weakness. Weaning from mechanical ventilation can be defined as the process of gradually withdrawing ventilatory support and liberating the patient from the endotracheal tube. The weaning process represents the 40-50% of the total duration of mechanical ventilation. Furthermore, a 26-42% rate of weaning failure has been reported after a single spontaneous breathing trial (SBT).It is well documented that weakness of the inspiratory muscles is a cause of weaning failure. Prolonged MV promotes diaphragmatic weakness due to both atrophy and contractile dysfunction. In addition, prolonged MV and weaning failure are indicators of poor prognosis. Prolonged ventilation increases the risk of complications, such as infections and critical illness neuromuscular syndromes Patients in the intensive care unit (ICU) who experience invasive mechanical ventilation for more than 72 h are susceptible to inspiratory muscle weakness. In patients invasively ventilated for longer than 7 days, this weakness manifests as impairments in both inspiratory muscle strength and endurance soon after ventilatory weaning. These impairments may contribute to elevated dyspnea in ICU patients both at rest and during exercise and thus hamper functional recovery. As ICU survivors often have poor levels of physical function and poor quality of life, interventions which improve strength and quality of life should be a priority for the healthcare team HYPOTHESES There is no difference between the effect of proprioceptive neuromuscular facilitation techniques versus Flow Trigger Sensitivity On Weaning Off Mechanical Ventilation

RESEARCH QUESTION:

Is there unique effect between Different proprioceptive neuromuscular facilitation techniques versus Flow Trigger Sensitivity On Weaning Off Mechanical Ventilation

ELIGIBILITY:
Inclusion Criteria:

1. Eighty four mechanically ventilated ICU patients under supervision; their age will be above 18 years old.
2. Mechanically ventilated due to type 1 or type 2 respiratory failures (RF) for at least 24 hours and Candidate for early extubation.
3. All patients are conscious and co-operative
4. All patients able to participate in training actively, weanable as regard to readiness weaning
5. All patients are hemodynamically stable.
6. Patient will be assigned in to three groups.
7. Presence of weaning criteria as defined in the European consensus conference in 2007, including sedation reduction, spontaneous breathing cycles, partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FiO2)150, absence of inotropes or vasopressors at high doses or increasing doses ( 1 mg/h),oxyhaemoglobin saturation (SaO2) 90% with FiO2 50% , positive end expiratory pressure (PEEP) 8 cmH2O,temperature is less than 38 ◦C.

Exclusion Criteria:

1. Hemodynamic or respiratory instability.
2. Condition that compromise weaning such as heart failure.
3. Condition that can prevent adequate performance of inspiratory muscle training such as neuropathy or myopathy.
4. Active hemorrhage and hemoptysis.
5. Large pneumothorax and pulmonary embolism.
6. Poor cognition and mentality.
7. Thoracic or abdominal surgery precluding the use of PNF exercises.
8. Rib fractures.
9. Current pregnancy.
10. Cardiac arrest with guarded neurological prognosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Maximum inspiratory pressure (MIP ) | 10 days
  Maximum inspiratory pressure (MIP ) is the "Negative inspiratory force" (NIF) , which is considered as a sensitive measure of respiratory muscle strength
Weaning success | 10 days
  weaning success is defined as extubation from mechanical ventilator without reintubation or death within 48 hours.

SECONDARY OUTCOMES:
Compliance (mL/cmH2O) | 10 days
  a. Static lung compliance
Respiratory rate | 10 days
  Respiratory Rate (RR) (breaths/min)
duration of mechanical ventilation | 10 days
  Duration of mechanical ventilation.
  .
Percentage of oxygen saturation | 10 days
  Percentage of oxygen saturation
Shallow rapid breathing index | 10 days
  Shallow rapid breathing index breath/min/ litter
Friction of inspired oxygen | 10 days
  Friction of inspired oxygen (FIO2)
Length of ICU stay | 10 days
  Length of ICU stay
Dynamic lung compliance | 10 days
  Dynamic lung compliance

CONTACTS AND LOCATIONS:
Overall Officials: Sherin Hassan Mehani, Professor of Physical Therapy, Principal Investigator — Faculty of Physical Therapy , Beni-Suef University
Locations (1):
- Beni-Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and summary of the results will be shared
Supporting Information: Study Protocol
Time Frame: Supporting information will be available after publishing the study till 12 months
Access Criteria: Supporting information will be available upon request from interested readers at the following E-mail :- sherinhassin@yahoo.com
URL: https://www.researchgate.net/search.Search.html?query=mehani+sherin&type=publication

REFERENCES:
- [Background] Ashtankar, A. P., Kazi, A., & Chordiya, S. (2019). Comparative effect of Proprioceptive Neuromuscular Facilitation (PNF) and chest physiotherapy with chest physiotherapy alone on SP02, heart rate, respiratory rate, & lung compliance in mechanically ventilated patient. J Pharm Sci Res, 11(10), 3514-8.
- [Background] Zwolinski T, Wujtewicz M, Szamotulska J, Sinoracki T, Waz P, Hansdorfer-Korzon R, Basinski A, Gosselink R. Feasibility of Chest Wall and Diaphragm Proprioceptive Neuromuscular Facilitation (PNF) Techniques in Mechanically Ventilated Patients. Int J Environ Res Public Health. 2022 Jan 15;19(2):960. doi: 10.3390/ijerph19020960. PMID 35055783
- [Background] de Souza RJP, Brandao DC, Martins JV, Fernandes J, Dornelas de Andrade A. Addition of proprioceptive neuromuscular facilitation to cardiorespiratory training in patients poststroke: study protocol for a randomized controlled trial. Trials. 2020 Feb 14;21(1):184. doi: 10.1186/s13063-019-3923-1. PMID 32059691
- [Background] Elbouhy, M. S., AbdelHalim, H. A., & Hashem, A. M. (2014). Effect of respiratory muscles training in weaning of mechanically ventilated COPD patients. Egyptian Journal of Chest Diseases and Tuberculosis, 63(3), 679-687.
- [Background] Ismail, O. A., El-Nahass, N. G., Abdeen, H. A., & Soliman, Y. (2021). Effect of Modifying Mechanical Ventilator Trigger Sensitivity on Arterial Blood Gases in ICU Patients. The Egyptian Journal of Hospital Medicine, 85(2), 3767-3771.